CLINICAL TRIAL: NCT03643445
Title: A Comparison of Motivation-Oriented Versus Psychoeducation-Oriented Day Hospital Treatment for Eating Disorders
Brief Title: Motivation-Oriented Versus Psychoeducation-Oriented Day Hospital Treatment for Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Collaborators: North York General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Jennifer Mills, Associate Professor, York University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160064
Record Dates: First submitted 2017-12-14; First posted 2018-08-22 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Motivational Interviewing; Psychoeducation
Keywords: motivational Interviewing; motivation; psychoeducation; psychoeducational-oriented treatment

STUDY DESIGN:
Intervention Model Description: Eating disorder participants will be randomly assigned either the motivation-oriented treatment condition or the psychoeducation-oriented treatment condition. Patients in both groups will receive the same care in terms of their hospital treatment and opportunities for interaction with the staff. The only difference will be that for ½ of participants, their treatment will be infused with motivation-oriented interventions. For the others, their interactions will be infused with psychoeducation-oriented interventions. All patients have interactions with an individual therapist at various time points in their hospital treatment. The points at which a patient meets with his or her individual therapist are as follows: at the orientation to the program, a 6-week check-in, and a 10-12 week check-in. As well, patients typically meet with their individual therapist whenever the treatment team determines that a patient may be struggling in the program and is at risk of premature drop-out.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (MI) Treatment (Experimental): Motivational interviewing is a psychotherapeutic stance aimed at helping patients in resolving ambivalence toward change and increasing their intrinsic motivation to engage in healthy behaviour choices. Patients assigned to these MI-trained therapists will be in the motivation-oriented condition. All individual meetings patients have with their therapist while they are in the program will entail sessions that are guided by MI principles. That is, revisiting patients' motivation to recover and overcoming obstacles to ambivalence or low motivation.
  Interventions: Behavioral: Motivational Orientated Treatment
- Psychoeducation-Oriented Treatment (Active Comparator): The psychoeducation-oriented treatment condition is intended to teach patients about the causes of eating disorders, the expected course of recovery, obstacles to recovery, and the importance of behavioural changes required for recovery from an eating disorder. Two staff members in the eating disorders program will deliver the psychoeducation-infused interventions, which are intended to be equivalent to treatment-as-usual in many eating disorder programs, but in a structured and standardized way, and with the use of the self-help manual. Psychoeducation is a very common intervention, often used as part of cognitive-behavioural treatment for eating disorders. The idea is that information about eating disorders and their health risks facilitates recovery and allows patients to "buy in" to treatment.
  Interventions: Behavioral: Psychoeducation-Oriented Treatment

INTERVENTIONS:
Behavioral: Motivational Orientated Treatment — The motivation-oriented treatment condition is intended to create a context for treatment that is patient-centered, non-judgmental, and will create a therapeutic environment wherein patients can make an informed decision around their goals for treatment and their willingness to commit to the behavioural changes required for recovery from an eating disorder. In general, MI is a psychotherapeutic stance aimed at helping patients in resolving ambivalence toward change and increasing their intrinsic motivation to engage in healthy behaviour choices.
  Arms: Motivational Interviewing (MI) Treatment
Behavioral: Psychoeducation-Oriented Treatment — The psychoeducation-oriented treatment condition is intended to teach patients about the causes of eating disorders, the expected course of recovery, obstacles to recovery, and the importance of behavioural changes required for recovery from an eating disorder. In this condition, in order to maximize the differences between groups, no attention will be given to discussing the patient's stage of change, their level of motivation, or their own personal values around recovery. Rather, emphasis during individual meetings with their therapist will be on the importance of symptom abstinence and normal eating.
  Arms: Psychoeducation-Oriented Treatment

SUMMARY:
1. Study Objectives To evaluate changes in general symptomatology in patients undergoing the day hospital eating disorders program at North York General Hospital and compare symptoms between treatment groups (motivation-oriented vs. psychoeducation-oriented).

   To determine treatment satisfaction ratings in patients undergoing the day hospital program and compare satisfaction between treatment groups.

   To evaluate the acceptability of patient-centered and motivation-oriented eating disorder treatment among patients.
2. Study Hypotheses:

Participants who receive motivation-oriented adjunctive treatment will experience larger improvements in eating disorder symptomatology 6 weeks into treatment, 10-12 weeks into treatment, and at discharge (compared to admission), and as compared to those receiving psychoeducation-oriented adjunctive treatment. Patients who receive motivation-oriented adjunctive treatment will report higher satisfaction with treatment, stronger feelings of motivation to recover, and will be more likely to complete the program as compared to those receiving psychoeducation-oriented adjunctive treatment.

DETAILED DESCRIPTION:
The Adult Eating Disorders Day Hospital Program at NYGH treats patients with a diagnosis of an eating disorder, including anorexia nervosa, bulimia nervosa, and other specified feeding and eating disorder. As with all intensive eating disorder treatment programs, relapse and drop-out are common occurrences. These outcomes are understood to occur when a patient is not ready to commit to the behavioural changes that are required for recovery, including normalized eating and abstinence from extreme food restriction, and bingeing and purging symptoms. Many patients struggle while they are in treatment for an eating disorder, demonstrating continued dietary restriction or urges to have symptoms like bingeing and purging.

The investigators are interested in examining whether modifications to the way in which the NYGH adult eating disorders program addresses motivation among patients will improve the quality, efficiency, and outcome of care. This study will compare two psychosocial adjunctive treatments during the standard hospital-based day treatment: one that focuses on patients' motivation to recover (motivational interviewing; MI) and the other that focuses on teaching patients about eating disorders and their associated risks (psychoeducation).

Informed by previous findings that a brief pre-treatment of MI can sometimes reduce treatment drop-out from intensive ED treatment, the current study aims to understand the effectiveness of motivation-oriented treatment for eating disorders. Based on previous research, if a patient is encouraged to reflect on and resolve obstacles to their readiness to change throughout the course of treatment, the researchers believe that objective treatment outcomes will improve alongside positive shifts in personal agency and confidence in one's ability to get better. Therefore, in addition to examining treatment completion and symptom improvement (as assessed by the standard questionnaires given to patients as part of program evaluation), the researchers will examine other psychological indicators of improvement that previous research has shown are important to consider in recovery, including treatment outcome expectancy (i.e., whether a patient feels confident that they can get better) as well as satisfaction with treatment.

The study will consist of two groups: patients will be randomly assigned to either motivation-oriented treatment or psychoeducation-oriented treatment. The researchers will include the fairly comprehensive package of outcome measures already administered to patients in this program to ensure that the researchers are looking at overall symptomatology in patients, as well as processes that could be expected to mediate outcome, such as patients' treatment outcome expectancies. The researchers will compare means on all measures between groups from pre-, mid- and end-of-treatment. The researchers believe that results from this study will add to the growing body of literature demonstrating the therapeutic benefit for motivation-oriented treatments for eating disorders and could assist the treatment team at NYGH and other hospitals with treatment planning.

ELIGIBILITY:
Inclusion Criteria:

1. Receiving treatment at NYGH in the Adult Eating Disorders Program
2. Over 17 years old
3. Able to speak and read English (minimum Grade 6 reading level)
4. Able to provide informed consent

Exclusion Criteria:

1. Not Applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Symptomatology | 8 weeks
  Standard questionnaire package that determines eating disorder symptomatology in eating disorder patients

SECONDARY OUTCOMES:
Self-ratings of motivation to recover | 8 weeks
  Measures readiness, confidence and importance of recovery
Self-ratings of Treatment Satisfaction | up to 24 weeks
  Measures treatment satisfaction
Completion of Program | up to 24 weeks
  Measures treatment program completion

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mills, Ph.D., Principal Investigator — North York General Hospital
Locations (1):
- North York General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Non-indentified individual participant data from outcome measures will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: approximately 6-7 months, post the study completion date, will the data be available.
Access Criteria: An independent external review board will be responsible for reviewing requests for data access.

REFERENCES:
- [Derived] Mills JS, Poulin LE, Kirsh G. Comparison of MI-oriented versus CBT-oriented adjunctive treatments: impacts on therapeutic alliance and patient engagement during hospital treatment for an eating disorder. J Eat Disord. 2023 Jun 20;11(1):98. doi: 10.1186/s40337-023-00818-8. PMID 37340439
- See also: Website of Principal Investigator — http://health.yorku.ca/health-profiles/index.php?mid=162289